CLINICAL TRIAL: NCT00792805
Title: A Phase III, 26-week Multicenter Randomized Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Indacaterol (150 and 300 µg Once Daily [od]) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Indacaterol in Adults (40 Years and Above) With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2333
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; indacaterol; long-acting β2-agonist; adults
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Indacaterol 150 μg (Experimental): Patients inhaled indacaterol 150 μg via a single-dose dry-powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM) for 26 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 µg
- Indacaterol 300 μg (Experimental): Patients inhaled indacaterol 300 μg via a single-dose dry-powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM) for 26 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg
- Placebo to indacaterol (Placebo Comparator): Patients inhaled placebo to indacaterol via a single-dose dry-powder inhaler (SDDPI) once daily (od) in the morning (between 8:00 and 11:00 AM) for 26 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 µg — Indacaterol was supplied in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Indacaterol 150 μg
Drug: Indacaterol 300 μg — Indacaterol was supplied in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Indacaterol 300 μg
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Placebo to indacaterol

SUMMARY:
This study evaluated the efficacy and safety of two doses of indacaterol in adults aged 40 or over with chronic obstructive pulmonary disease (COPD) in China and in two other countries.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years
* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate to severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2007) and:

  1. Smoking history of at least 10 pack years
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

* Patients who have received systemic corticosteroids for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period
* Patients requiring long-term oxygen therapy (> 15 hours a day) for chronic hypoxemia
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Any patient with active cancer or a history of cancer with less than 5 years disease-free survival time
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at screening is prolonged
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period
* Patients unable to successfully use a dry powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Australia (3):
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Clayton
  - Novartis Investigative Site, Daw Park
- China (10):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Changsha
  - Novartis Investigative Site, Chongqing
  - Novartis Investigator Site, Fuzhou
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shandong
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenyang
  - Novartis Investigative Site, Shijiazhuang
  - Novartis Investigative Site, Xi'an
- India (2):
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Trivandrum

REFERENCES:
- [Derived] Yao W, Wang C, Zhong N, Han X, Wu C, Yan X, Chen P, Yang W, Henley M, Kramer B. Effect of once-daily indacaterol in a predominantly Chinese population with chronic obstructive pulmonary disease: a 26-week Asia-Pacific study. Respirology. 2014 Feb;19(2):231-238. doi: 10.1111/resp.12211. Epub 2014 Jan 3. PMID 24383720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo to Indacaterol
Started | 188 | 188 | 187
Exposed to Study Medication or Placebo | 187 (One patient in this group did not receive any study treatment.) | 188 | 186 (One patient in this group did not receive any study treatment.)
Completed | 166 | 162 | 154
Not Completed | 22 | 26 | 33
Not completed — Adverse Event | 12 | 10 | 10
Not completed — Subject withdrew consent | 5 | 6 | 5
Not completed — Administrative problems | 2 | 0 | 4
Not completed — Abnormal test procedure result(s) | 1 | 2 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 6 | 6
Not completed — Lost to Follow-up | 1 | 1 | 6
Not completed — Abnormal laboratory value(s) | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo to Indacaterol | Total
Number analyzed (Participants) | 187 | 188 | 186 | 561
Age Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.01) | 65.5 (8.86) | 64.6 (9.30) | 65.4 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 13 | 32
  Male | 175 | 181 | 173 | 529

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12 + 1 Day, Day 85
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1 and FEV1 pre-dose and 10-15 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Week 12 + 1 day, Day 85
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug. Last observation carried forward (LOCF) was utilized to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo to Indacaterol
Number analyzed (Participants) | 176 | 178 | 171
Liters | 1.32 (0.024) | 1.29 (0.024) | 1.17 (0.024)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 26)
Description: Safety population: All patients who received at least 1 dose of study drug.
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 12/187 | 12/188 | 15/186
Other Adverse Events (participants affected / at risk) | 38/187 | 50/188 | 47/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=187) | Indacaterol 300 μg (N=188) | Placebo to Indacaterol (N=186)
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Eye oedema (Eye disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=187) | Indacaterol 300 μg (N=188) | Placebo to Indacaterol (N=186)
Nasopharyngitis (Infections and infestations) | 16 | 14 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 13 | 16
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 29 | 35 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.